CLINICAL TRIAL: NCT07041242
Title: Outcomes and Complication Rates of Anterior Cruciate Ligament Reconstruction Using the "Over-the-top" Technique Combined With Lateral Extra-articular Tenodesis in Patients Over 50 Years Old, Compared With a Control Group of Patients Under 30
Acronym: ACL_50_YO
Status: Recruiting | Type: Observational
Sponsor: Stefano Zaffagnini (Other)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: ACL_50_YO
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: ACL; LET; Hamstring Muscles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- over 50
  Interventions: Procedure: ligament reconstruction using the single-bundle "over-the-top" technique
- under 30
  Interventions: Procedure: ligament reconstruction using the single-bundle "over-the-top" technique

INTERVENTIONS:
Procedure: ligament reconstruction using the single-bundle "over-the-top" technique — Patients who have undergone anterior cruciate ligament reconstruction using the single-bundle "over-the-top" technique with gracilis and semitendinosus tendons, combined with a lateral extra-articular tenodesis, will be enrolled

SUMMARY:
The anterior cruciate ligament (ACL) is one of the main stabilizers of the knee, and its injury is among the most common soft tissue injuries of the knee. Surgical reconstruction of the ACL can be performed using various techniques and different types of tissue grafts, including both autografts and allografts.

Although ACL reconstruction is a widely performed surgical procedure in young and physically active individuals-typically patients under 30 years of age-to promote return to sports and prevent early onset of osteoarthritic degeneration, the surgical approach has historically been less common in patients over the age of 50. This is largely due to the lower functional demands typically observed in older patients.

However, with increasing life expectancy and a corresponding rise in functional demands among older individuals, the surgical approach to ACL reconstruction has been progressively reconsidered in the over-50 population. Several recent studies have aimed to evaluate the outcomes of ACL reconstruction in older adults, showing promising results in terms of both recurrence rates and complication rates.

At the II Clinic of the Rizzoli Orthopaedic Institute, under the direction of Professor Zaffagnini, the preferred technique for ACL reconstruction is the "single-bundle over-the-top technique using gracilis and semitendinosus tendons, combined with a lateral extra-articular tenodesis (LET)." LET is an additional surgical step performed alongside ACL reconstruction, which has shown excellent results, especially in young patients at high risk of reinjury. Specifically, clinical data have shown that adding LET to ACL reconstruction can reduce the failure rate by approximately 30%, significantly improve knee stability, and enable a faster return to sports-all without increasing the rate of complications compared to the standard isolated ACL reconstruction technique.

Given these encouraging results in terms of safety and reduced failure rates, the combined ACL + LET procedure has historically been used at the Rizzoli Orthopaedic Institute for all patients, including those over 50 years of age.

The consistent use of this technique allows for the creation of a homogeneous patient cohort, all treated with the same surgical approach. This also enables the formation of two comparable patient groups-one over 50 and one under 30-both treated with the same technique, allowing for a meaningful comparison of primary and secondary endpoints.

While several studies have aimed to compare ACL reconstruction outcomes in older populations with those in younger cohorts, to date, there are no studies in the literature that specifically assess the outcomes and complication rates of ACL reconstruction using the over-the-top technique combined with LET in patients over 50, and compare them with those of younger patients undergoing the same surgical procedure.

Given the growing demand for ACL reconstruction in older patients, we believe it is important to evaluate outcomes in patients over 50 and compare them with a younger cohort, to determine whether the over-the-top + LET technique may be a valid therapeutic option not only for young patients but also for older adults.

Of particular interest is the assessment of the reduced risk of failure and complication rate of the ACL + LET technique performed in over-50 patients, to determine whether the excellent clinical outcomes observed in younger individuals are also confirmed in an older population.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on between 2007 and 2023 who were over 50 years old at the time of surgery (study group) and patients under 30 years old at the time of surgery (control group).
* Patients who underwent ACL reconstruction using the gracilis and semitendinosus tendons with the over-the-top + LET technique.
* Patients of both male and female sex.
* Patients who have provided consent to participate in the study.

Exclusion Criteria:

* Previous surgery on the same limb (meniscectomy, prior ACL reconstruction, surgically treated fractures, osteotomies, meniscal transplants).
* Concomitant surgery on the same limb (osteotomies, meniscal transplants).
* Surgical technique different from the over-the-top with LET using autologous gracilis and semitendinosus tendons.
* Other concomitant ligament injuries requiring surgical treatment.
* Patients younger than 18 years at the time of surgery (minors) or patients aged between 30 and 50 years at the time of surgery.
* Patients who have not provided informed consent.
* Patients with a follow-up period shorter than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from both male and female subjects over 50 years of age at the time of surgery (study group), and adult patients, also both male and female, aged between 18 and 30 years at the time of surgery (control group), who underwent surgical treatment at the II Clinic of the Rizzoli Orthopaedic Institute by means of single-bundle "over-the-top" anterior cruciate ligament reconstruction using the gracilis and semitendinosus tendons, combined with lateral extra-articular tenodesis.
  Only patients at least 2 years post-surgery will be enrolled. Patients will be recruited evenly and progressively to ensure proper matching of the two groups with respect to patient characteristics. For each patient over 50 included in the study, a patient under 30 with similar characteristics (total follow-up duration, sex, concomitant meniscal injuries at the time of surgery) will be included to guarantee a balanced comparison between the two patient cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Complications | 2 years
  Any complications and subsequent procedures will be documented and recorded in the Case Report Form (CRF). The staff responsible for distributing and collecting the questionnaires will assign an identification code on the front page of each questionnaire in order to safeguard the privacy of the study participants.

SECONDARY OUTCOMES:
Lysholm Knee Score | 2 years
  It is a validated measurement scale that assesses knee functionality through 8 items, which help determine the condition of the knee in response to the functional demands of daily activities. This evaluation form is used to assess surgical outcomes in patients who have undergone surgery for ligament or meniscal injuries of the knee.
  The final score is obtained by summing the individual item scores and ranges from 0 to 100. The scores are classified into subgroups as follows:
  * Excellent (95-100)
  * Good (84-94)
  * Fair (65-83)
  * Poor (<64)
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 2 years
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is used to assess both short-term and long-term outcomes in patients following a knee injury. The self-administered KOOS evaluates five domains: pain, symptoms, activities of daily living, sport and recreational function, and knee-related quality of life.
  KOOS meets core standards for outcome measures and can be used to monitor the progression of knee injury and the effectiveness of treatment. The KOOS questionnaire includes five dimensions relevant to patients: pain, symptoms, daily living activities, sports and recreational activities, and quality of life.
  Each dimension is assessed separately using a five-point Likert scale, ranging from 0 (no problems) to 4 (extreme problems).
Visual Analog Scale (VAS) | 2 years
  The Visual Analog Scale (VAS) is a one-dimensional, quantitative 10-point numerical scale used to assess pain. Patients are asked to select the number that best describes the intensity of their pain at that specific moment, with 0 indicating no pain and 10 representing the worst possible pain.
  This scale will also be used to assess both preoperative and postoperative pain in the lateral compartment of the knee. The data will help evaluate the onset of pain following surgery, specifically in the area where metal staples are placed for graft fixation during the lateral extra-articular tenodesis procedure.
  Pain reported in the lateral femorotibial compartment with a VAS score greater than 2 will be considered indicative of the presence of lateral compartment pain, while a score of 2 or less will be considered as the absence of pain in that area.
Tegner Score | 2 years
  This scale is used to estimate an individual's level of physical activity, with scores ranging from 0 to 10. A score of 0 represents "disability," while a score of 10 indicates participation in competitive sports, such as national or international level football. The Tegner Score is one of the most commonly used tools to define the activity level of patients with knee disorders.
  In this study, the Tegner Score will be completed directly by the investigator through an interview with the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy